CLINICAL TRIAL: NCT02333942
Title: A Non-Blinded, Non-Significant Risk Study With a Non-Invasive, Passive Pressure Wave Method of Diagnosing Brain Pathologies to Develop a Diagnostic Algorithm for Alzheimer Disease and Other Dementias.
Brief Title: Dementia Signal Development Study of Nautilus NeuroWave TM for the Detection of Dementia
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 082189
Record Dates: First submitted 2014-12-09; First posted 2015-01-08 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Frontotemporal Lobar Degeneration; Memory Disorders
Keywords: Aging; Diagnostic Equipment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Frontotemporal Lobar Degeneration; Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Alzheimer's Disease: Nautilus NeuroWaveTM System'
  Interventions: Device: Nautilus NeuroWaveTM System
- Mild Cognitive Impairment: Nautilus NeuroWaveTM System'
  Interventions: Device: Nautilus NeuroWaveTM System
- Frontotemporal Lobar Degeneration: Nautilus NeuroWaveTM System'
  Interventions: Device: Nautilus NeuroWaveTM System
- Age-Matched Controls: Nautilus NeuroWaveTM System'
  Interventions: Device: Nautilus NeuroWaveTM System

INTERVENTIONS:
Device: Nautilus NeuroWaveTM System — A noninvasive device to detect dementia utilizing headset and sensors

SUMMARY:
This study is being performed to generate data regarding brain vibration /oscillation differences between individuals with dementia and normal controls. The purpose of this study is to compare signal patterns generated from the impact on the scalp from these brain oscillation patterns from individuals with Alzheimer's disease, Frontotemporal Lobar Degeneration, Mild Cognitive Impairment and Age-Matched Normal Controls.

DETAILED DESCRIPTION:
This is a non-blinded study in subjects who present to the UCSF Memory and Aging Clinic (MAC) with neurodegenerative disease and cognitive dysfunction. The primary objective of this non-significant risk study is signature development. The goal is to develop a signal algorithm using the Nautilus NeuroWaveTM for dementia. This is accomplished by analyzing and processing Nautilus NeuroWave recordings from a patient with confirmed dementia. All subjects will be enrolled until recordings are obtained from at least 10 of each of the following subject cohorts: Moderate or Severe Frontotemporal Lobar Degeneration (FTDL), Alzheimer's Disease, Mild Cognitive Impairment (MCI) and Age Matched Normal Controls.

As this study is a feasibility study intended to determine whether the Nautilus NeuroWave is able to generate distinctive signals correlated with dementia, statistical analysis will not be required. Similarly, the study has not been powered to attain any particular level of statistical significance. Subsequent studies will measure sensitivity and specificity of any resulting dementia signal pattern generated by this study. These future studies will be subject to statistical analysis.

The Jan Medical Nautilus NeuroWaveTM (NNW) is a non-invasive device designed to evaluate brain oscillation patterns or the brain's pulse, generated by cardiac cycle induced intracranial blood flow. The objective of the evaluation is to determine whether the oscillation pattern is normal, whether it has been disrupted, and, if disrupted, what particular disruption pattern is evident. Various cerebral pathologies studied to date with the NNW demonstrate distinct disruption patterns. These pathologies include vasospasm, concussion and arterio-venous malformation (AVM). The objective of this study is to evaluate the brain oscillation patterns from subjects with MCI, Frontotemporal dementia, AD and from a small cohort of age matched normal controls and determine whether they exhibit pattern disruption and, if so, to quantify and categorize the distinct disruption patterns. How the Nautilus NeuroWave accomplishes this is explained later in the device description section of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older
2. Have undergone some neurologic imaging
3. Age match normal subjects and subjects with symptoms consistent with MCI, FTLD or Alzheimer's disease
4. Able to understand and provide signed informed consent, or have a legally authorized representative willing to provide informed consent on subject's behalf

Exclusion Criteria:

1. Psychologically unstable and not able to cooperate
2. Not suitable for participation in this study in the opinion of the PI
3. Patients with history of other cerebral pathologies including, head trauma or prior ICH

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Alzheimer's Disease, Frontotemporal Lobar Degeneration, Mild Cognitive Impairment, and Age-Matched Controls.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity as a diagnostic aid in detecting Dementia (identified signatures as compared with the clinical assessment made by the PI) | one year
  Efficacy at identifying Dementia through identified signatures as compared with the clinical assessment made by the PI and any objective measures the PI uses to arrive at assessment.
Specificity as a diagnostic aid in detecting Dementia (Rate of false positives as compared with the clinical assessment made by the PI) | one year
  Rate of false positives as compared with the clinical assessment made by the PI and any objective measures the PI uses to arrive as assessment.

SECONDARY OUTCOMES:
Sensitivity and specificity measures for MCI and Alzheimer's disease (Efficacy and rate of false positives as compared with the clinical assessment made by the PI) | one year
  Efficacy and rate of false positives as compared with the clinical assessment made by the PI and any objective measures the PI uses to arrive as assessment.
Sensitivity and specificity measures between MCI and FTDL. (distinguish between MCI and FTDL using efficacy and rate of false positives from the identified signatures as compared with the clinical assessment made by the PI) | one year
  To distinguish between MCI and FTDL using efficacy and rate of false positives from the identified signatures as compared with the clinical assessment made by the PI and any objective measures the PI uses to arrive as assessment.
Sensitivity and specificity measures between FTDL and Alzheimer's disease (distinguish between FTLD and Alzheimer's disease using efficacy and rate of false positives from the identified signatures as compared with the clinical assessment made by the PI) | one year
  To distinguish between FTLD and Alzheimer's disease using efficacy and rate of false positives from the identified signatures as compared with the clinical assessment made by the PI and any objective measures the PI uses to arrive as assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Kao, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Californa San Francisco, San Francisco, California, United States